CLINICAL TRIAL: NCT02847624
Title: Post-Marketing Surveillance Study of Tolvaptan in Patients With ADPKD in Japan
Brief Title: Post-Marketing Surveillance Study of Tolvaptan in Patients With ADPKD
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 15600-003
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ADPKD
  Interventions: Drug: tolvaptan

INTERVENTIONS:
Drug: tolvaptan

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of tolvaptan in patients with autosomal dominant polycystic kidney disease (ADPKD) in the real world clinical setting in Japan.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed ADPKD
* total kidney volume of 750 or more

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: medical institutes all over Japan
Sampling Method: Non-Probability Sample
Enrollment: 1802 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Fukuta, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Otsuka Pharmaceutical Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mochizuki T, Muto S, Suzue K, Komaniwa S, Tanaka T, Fukuta Y, Yamashige Y. Safety and efficacy of tolvaptan in real-world Japanese patients with autosomal dominant polycystic kidney disease: final results of SLOW-PKD surveillance. Clin Exp Nephrol. 2025 Jun;29(6):807-817. doi: 10.1007/s10157-025-02634-7. Epub 2025 Feb 14. PMID 39953249

RESULTS

PARTICIPANT FLOW:
Groups:
- ADPKD: Patients with a diagnosis of ADPKD, a TKV of more than 750 mL, and an annual TKVslope increase of more than 5% as measured by magnetic resonance imaging (MRI), computed tomographic (CT) scanning, or ultrasound were included.
Period: Overall Study
Arm/Group | ADPKD
Started | 1802
Completed | 1672
Not Completed | 130
Not completed — Lost to Follow-up | 28
Not completed — Protocol Violation | 98
Not completed — Case report failures | 4

BASELINE CHARACTERISTICS:
Arm/Group | ADPKD
Number analyzed (Participants) | 1672
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 1479
  >=65 years | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 805
  Male | 867
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1672
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 1672
Weight [Mean (Standard Deviation); unit: kg] | 64.2 (12.7)
Complication [Count of Participants; unit: Participants]
  Hypertension | 1447
  Diabetes | 74
  Hyperlipidaemia | 460
  Hyperuricaemia | 746
  Liver disease(Cystic liver) | 739
  Liver disease(others) | 54
  Pancreatic cysts | 19
  Cerebral aneurysm | 161
  Kidney disease | 254
  Urinary calculus | 36
  Cyst infection | 26
  Urinary tract infection | 7
Predisposition to hypersensitivity [Count of Participants; unit: Participants]
  None | 1411
  Medicine | 49
  Foods | 39
  Others | 144
  Missing | 56
History of drug adverse reactions [Count of Participants; unit: Participants]
  None | 1536
  Any | 91
  Missing | 45

OUTCOME MEASURES:

1. Primary Outcome: Estimated Slope of Total Kidney Volume During Pre-administration and Administration
Description: Total Kidney Volume (TKV) was used as a biomarker to assess the progression of ADPKD. TKV was measured at each participating site based on imaging obtained via ultrasound, CT, or MRI.
  The Estimated Slope pre-administration was calculated for subjects who had TKV measurements both prior to and on the day of Tolvaptan initiation (baseline). The rate of change in TKV from the pre-treatment measurement date to the baseline was used to determine the Estimated Slope.
  Since the date of initiating tolvaptan administration is considered the start date of the study, the kidney volume measured prior to administration falls outside the study period (i.e., it is a value from before the study start date).
  The Estimated Slope during-treatment was calculated for subjects who had bilateral TKV measurements at baseline and during the treatment period. The rate of change in TKV from baseline to the measurement date during treatment was used to determine the Estimated Slope.
Time Frame: Pre-administration: From the first pre-treatment measurement (up to 12.5 years prior) to the start of tolvaptan. During-treatment: From the start of tolvaptan to the final follow-up (up to 8.0 years later).
Population: Pre-administration: Estimated slope was calculated in cases with both pre-treatment and baseline TKV data.
  During-treatment: Estimated slope was calculated in cases with both baseline and on-treatment TKV data.
  Because this study used real-world clinical data, not all patients had both sets of measurements required for either group. As a result, the number of cases included in the pre-administration and during-treatment groups was smaller than the total of 1,672 cases analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: %/year
Groups:
- ADPKD: Patients with a diagnosis of ADPKD, a TKV of more than 750 mL, and an annual TKV slope increase of more than 5% as measured by magnetic resonance imaging (MRI), computed tomographic (CT) scanning, or ultrasound were included.
Arm/Group | ADPKD
Number analyzed (Participants) | 1672
%/year
  Pre-administration: number analyzed (Participants) | 826
  Pre-administration | 6.7517 (0.2183)
  During administration: number analyzed (Participants) | 1369
  During administration | 3.6811 (0.9514)

2. Secondary Outcome: The Number of Cases in Which ALT Never Exceeded Three Times the Upper Limit of Normal (30 IU/L)
Description: Among cases included in the safety analysis, we counted and listed the number of patients whose ALT levels increased after starting tolvaptan but never exceeded three times the upper limit of normal (30 IU/L) at a specific time point (day) during treatment.
  Cases in which Tolvaptan treatment was discontinued were considered as dropouts on the day of discontinuation.
  The number of participants analyzed in each row of the data table is the same as the Overall Number of Participants Analyzed (n=1,672)
Time Frame: From the date of Tolvaptan initiation to the earlier of either the date when ALT reached three times the upper limit of normal or the date of Tolvaptan discontinuation (up to 2789 days).
Population: Safety analysis population (n = 1,672)
Measure: Number; unit: participants
Arm/Group | ADPKD
Number analyzed (Participants) | 1672
participants
  Baseline | 1672
  500 days | 1210
  1000 days | 1007
  1500 days | 706
  2000 days | 402
  2500 days | 47
  3000 days | 0

3. Secondary Outcome: The Number of Cases in Which AST Never Exceeded Three Times the Upper Limit of Normal (30 IU/L)
Description: Among cases included in the safety analysis, we counted and listed the number of patients whose AST levels increased after starting tolvaptan but never exceeded three times the upper limit of normal (30 IU/L) at a specific time point (day) during treatment.
  Cases in which Tolvaptan treatment was discontinued were considered as dropouts on the day of discontinuation.
  The number of participants analyzed in each row of the data table is the same as the Overall Number of Participants Analyzed (n=1,672)
Time Frame: From the date of Tolvaptan initiation to the earlier of either the date when AST reached three times the upper limit of normal or the date of Tolvaptan discontinuation (up to 2789 days).
Population: Safety analysis population (n = 1,672)
Measure: Number; unit: participants
Arm/Group | ADPKD
Number analyzed (Participants) | 1672
participants
  Baseline | 1672
  500 days | 1232
  1000 days | 1027
  1500 days | 715
  2000 days | 413
  2500 days | 47
  3000 days | 0

4. Other Pre Specified Outcome: Estimated Slope of Estimated Glomerular Filtration Rate (e-GFR) During Pre-administration and Administration
Description: e-GFR was used as a biomarker to evaluate ADPKD progression. Values recorded in the CRF were prioritized; if unavailable, e-GFR was calculated using serum creatinine levels with a gender-specific formula.
  Male:
  e-GFR=194×(serum creatinine (mg/dL))^-1.094 ×(age)^-0.287
  Female:
  e-GFR=[194×(serum creatinine (mg/dL))^-1.094 ×(age)^-0.287]×0.739 The pre-treatment Estimated Slope was determined for subjects with e-GFR data both before and at the start of tolvaptan administration (baseline). Since the date of initiating tolvaptan administration is considered the start date of the study, the e-GFR measured prior to administration falls outside the study period.
  The during-treatment Estimated Slope was calculated for subjects with e-GFR measurements at baseline and during treatment, based on the rate of change from baseline to follow-up.
Time Frame: Pre-administration: From the first pre-treatment measurement (up to 10 years prior) to the start of tolvaptan. During-treatment: From the start of tolvaptan to the final follow-up (up to 8.0 years later).
Population: Pre-administration: Estimated slope was calculated in cases with both pre-treatment and baseline e-GFR data.
  During-treatment: Estimated slope was calculated in cases with both baseline and on-treatment e-GFR data.
  Because this study used real-world clinical data, not all patients had both sets of measurements required for either group. As a result, the number of cases included in the pre-administration and during-treatment groups was smaller than the total of 1672 cases analyzed for efficacy.
Measure: Mean (Standard Error); unit: %/year
Arm/Group | ADPKD
Number analyzed (Participants) | 1672
%/year
  Pre-administration: number analyzed (Participants) | 1034
  Pre-administration | -3.6272 (0.3572)
  During-treatment: number analyzed (Participants) | 1626
  During-treatment | -3.2561 (0.0552)

5. Other Pre Specified Outcome: The Number and Percentage of Adverse Events Observed in Patients Aged 65 Years and Older
Description: The incidence rates of Adverse Drug Reactions(ADRs) were calculated for 192 elderly patients aged 65 years and older, and compared with those in non-elderly patients under 65 years of age.
Time Frame: Adverse events were collected during the period from the start date to the end date of tolvaptan administration for each case (max. 8 years).
Population: Elderly patients: Aged 65 years and older Non-elderly patients: Aged under 65 years
Measure: Count of Participants; unit: Participants
Arm/Group | ADPKD
Number analyzed (Participants) | 1672
Participants
  Elderly patients: number analyzed (Participants) | 192
  Elderly patients | 87
  Non-elderly patients: number analyzed (Participants) | 1480
  Non-elderly patients | 690

6. Other Pre Specified Outcome: Safety in Patients With Advanced ADPKD
Description: Adverse events were summarized in patients with advanced ADPKD who had their creatinine clearance measured at the start of tolvaptan treatment.
  Patients with advanced ADPKD were defined as those with a pre-treatment creatinine clearance of less than 60 mL/min. The incidence rates of Adverse Drug Reactions(ADRs) were calculated for 752 patients with creatinine clearance <60 mL/min, 261 patients with clearance between 60 and <80 mL/min, and 331 patients with clearance ≥80 mL/min, and the rates were compared across the creatinine clearance groups.
Time Frame: as for outcome 5
Population: The study cases were divided into the following three groups based on creatinine clearance before administration, and the incidence rate of ADRs was calculated for each group: less than 60 mL/min, 60 to less than 80 mL/min, and 80 mL/min or more.
Measure: Count of Participants; unit: Participants
Arm/Group | ADPKD
Number analyzed (Participants) | 1344
Participants
  creatinine clearance <60 mL/min: number analyzed (Participants) | 752
  creatinine clearance <60 mL/min | 346
  creatinine clearance between 60 and <80 mL/min: number analyzed (Participants) | 261
  creatinine clearance between 60 and <80 mL/min | 129
  creatinine clearance ≥80 mL/min: number analyzed (Participants) | 331
  creatinine clearance ≥80 mL/min | 157

7. Other Pre Specified Outcome: Safety of Long-term Treatment for ADPKD
Description: In the clinical trials conducted prior to approval, there were no cases in which Samsca was administered continuously for more than three years. In this post-marketing surveillance, cases exceeding the three-year (36-month) treatment period of the pre-approval clinical trials were classified as long-term treatment cases. The safety of long-term treatment was evaluated based on the incidence rate of adverse drug reactions (ADRs) according to the timing of their onset.
Time Frame: as for outcome 5
Population: The incidence rate of ADRs was calculated for each time interval from the start of administration. Cases exceeding 36 months were classified as long-term treatment. In cases where the same ADR occurred multiple times in the same patient, all occurrences were included in the calculation.
Measure: Count of Participants; unit: Participants
Arm/Group | ADPKD
Number analyzed (Participants) | 1672
Participants
  ≤7 days: number analyzed (Participants) | 1667
  ≤7 days | 201
  8-14 days: number analyzed (Participants) | 1656
  8-14 days | 45
  15-21 days: number analyzed (Participants) | 1649
  15-21 days | 45
  >21 days to ≤3 months: number analyzed (Participants) | 1639
  >21 days to ≤3 months | 165
  >3 to ≤6 months: number analyzed (Participants) | 1587
  >3 to ≤6 months | 174
  >6 to ≤9 months: number analyzed (Participants) | 1484
  >6 to ≤9 months | 129
  >9 to ≤12 months: number analyzed (Participants) | 1422
  >9 to ≤12 months | 78
  >12 to ≤24 months: number analyzed (Participants) | 1387
  >12 to ≤24 months | 129
  >24 to ≤36 months: number analyzed (Participants) | 1175
  >24 to ≤36 months | 120
  >36 to ≤48 months: number analyzed (Participants) | 968
  >36 to ≤48 months | 56
  >48 to ≤60 months: number analyzed (Participants) | 772
  >48 to ≤60 months | 40
  >60 to ≤72 months: number analyzed (Participants) | 470
  >60 to ≤72 months | 30
  >72 to ≤84 months: number analyzed (Participants) | 77
  >72 to ≤84 months | 3
  >84 months: number analyzed (Participants) | 10
  >84 months | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the period from the start date to the end date of tolvaptan administration for each case (max. 8 years).
Description: The adverse events (if any occurred), onset date, seriousness, reason to have judge the event as serious (in case of serious), outcome, date of outcome judgement, causality to tolvaptan, other possible causal factors, and treatment for adverse events during the observation period were recorded. Seriousness was determined by the physicians.
Arm/Group | ADPKD
All-Cause Mortality (participants affected / at risk) | 21/1672
Serious Adverse Events (participants affected / at risk) | 253/1672
Other Adverse Events (participants affected / at risk) | 1086/1672
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADPKD (N=1672)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 2 (2)
Chronic Heart Failure (Cardiac disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 3 (3)
Colonic polyps (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 4 (4)
Death (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Hemorrhagic cyst (General disorders) | 3 (3)
Peripheral edema (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Drug-induced Liver Injury (Hepatobiliary disorders) | 3 (3)
Liver Cysts (Hepatobiliary disorders) | 2 (2)
Liver Damage (Hepatobiliary disorders) | 8 (8)
Liver Dysfunction (Hepatobiliary disorders) | 14 (14)
Appendicitis (Infections and infestations) | 3 (3)
Cellulitis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Infectious Cyst (Infections and infestations) | 13 (13)
Liver Cyst Infection (Infections and infestations) | 8 (8)
Peritonitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 4 (4)
Renal Cyst Infection (Infections and infestations) | 32 (32)
Sepsis (Infections and infestations) | 3 (3)
Septic Shock (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Scar hernia (Injury, poisoning and procedural complications) | 2 (2)
Subdural hematoma (Injury, poisoning and procedural complications) | 4 (4)
Increase in Blood Creatinine (Investigations) | 2 (2)
Increase in Blood Osmotic Pressure (Investigations) | 2 (2)
Increase in C-Reactive Protein (Investigations) | 2 (2)
Increase in Liver Enzymes (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Loss of appetite (Metabolism and nutrition disorders) | 2 (2)
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Liver Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Malignant Neoplasm of the Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Altered state of consciousness (Nervous system disorders) | 2 (2)
Cerebral hemorrhage (Nervous system disorders) | 3 (3)
Cerebral infarction (Nervous system disorders) | 3 (3)
Intracranial aneurysm (Nervous system disorders) | 5 (5)
Putaminal hemorrhage (Nervous system disorders) | 2 (2)
Subarachnoid hemorrhage (Nervous system disorders) | 11 (11)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Chronic Kidney Disease (Renal and urinary disorders) | 6 (6)
End-Stage Renal Disease (Renal and urinary disorders) | 4 (4)
Hematuria (Renal and urinary disorders) | 2 (2)
Renal Cyst Hemorrhage (Renal and urinary disorders) | 15 (15)
Renal Dysfunction (Renal and urinary disorders) | 11 (11)
Renal Failure (Renal and urinary disorders) | 15 (15)
Ureteral Calculi (Renal and urinary disorders) | 5 (5)
Prostatitis (Reproductive system and breast disorders) | 2 (2)
Severe menstrual bleeding (Reproductive system and breast disorders) | 2 (2)
Aortic Dissection (Vascular disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADPKD (N=1672)
Pharyngitis (Infections and infestations) | 46 (46)
Renal Cyst Infection (Infections and infestations) | 45 (45)
Hyperkalemia (Metabolism and nutrition disorders) | 61 (61)
Hypernatremia (Metabolism and nutrition disorders) | 93 (93)
Hyperuricemia (Metabolism and nutrition disorders) | 177 (177)
Hypertension (Vascular disorders) | 50 (50)
Constipation (Gastrointestinal disorders) | 35 (35)
Liver Function Disorder (Hepatobiliary disorders) | 178 (178)
Liver Disorder (Hepatobiliary disorders) | 59 (59)
Back Pain (Musculoskeletal and connective tissue disorders) | 44 (44)
Renal Failure (Renal and urinary disorders) | 34 (34)
Renal Dysfunction (Renal and urinary disorders) | 106 (106)
Thirst (General disorders) | 135 (135)
Increased Blood Creatine Phosphokinase (Investigations) | 43 (43)
Increased Blood Creatinine (Investigations) | 36 (36)
Increased Gamma-Glutamyltransferase (Investigations) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT02847624/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT02847624/SAP_001.pdf